CLINICAL TRIAL: NCT03187353
Title: Multi-Modal Imaging of Psychostimulant Effects on Executive Function Post-RRSO
Brief Title: IMProving Executive Function Study
Acronym: IMPRES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 826981
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Impairment; RRSO
Keywords: Cognitive complaints; RRSO; Oophorectomy; Memory; Cognition; Early menopause
MeSH Terms: conditions — Cognitive Dysfunction; Primary Ovarian Insufficiency | interventions — Lisdexamfetamine Dimesylate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lisdexamfetamine, then Placebo (Experimental): Participants will have a 50% chance of first receiving the active study medication. They will begin at 20 mg/d and will increase up to 60 mg/d after 4 weeks, if well tolerated. Total time on the study drug is up to 6 weeks. After a washout period of 2 weeks they will begin with 1 sugar pill and will increase up to 3 pills after 4 weeks. Maximum time for taking the placebo is 6 weeks.
  Interventions: Drug: Lisdexamfetamine; Drug: Placebo oral capsule
- Placebo, then Lisdexamfetamine (Experimental): Participants will have a 50% chance of first receiving the placebo, beginning with 1 sugar pill and increasing up to 3 pills after 4 weeks. Maximum time for taking the placebo is 6 weeks. After a washout period of 2 weeks, they will begin active study medication at 20 mg/d and will increase up to 60 mg/d after 4 weeks, if well tolerated. Total time on the study drug is up to 6 weeks.
  Interventions: Drug: Lisdexamfetamine; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Lisdexamfetamine — Stimulant medications are used to reduce interruptive behavior, fidgeting, and other hyperactive symptoms, as well as help a person finish tasks and improve his or her relationships for adults who have ADHD. Please note that the FDA has not approved the use of Vyvanse® for the treatment of memory and concentration difficulties related to medically induced menopause.
  Other Names: Vyvanse
Drug: Placebo oral capsule — The placebo capsule will be filled with microcellulose.
  Other Names: sugar pill

SUMMARY:
This is a double-blind, placebo-controlled, crossover study testing whether Vyvanse (lisdexamfetamine; LDX) improves executive functioning (EF) in 100 postmenopausal women who report onset of EF difficulties after oophorectomy. This study involves magnetic resonance imaging (MRI) to see how LDX affects brain chemistry while undergoing two 6-week trials of the study drug and placebo capsules.

UPDATE: We have recently updated this protocol (09/2020) to offer a remote version of the study that can be completed entirely from the participant's home. This alternate version of the study eliminates travel, the MRI, and blood draws.

DETAILED DESCRIPTION:
Following a medically induced menopause, many women report difficulty in remembering things, focusing and concentrating. The purpose of this study is to examine the effects of a stimulant medication called Vyvanse® (lisdexamfetamine; LDX) on executive functioning, such as attention, processing, organization, and memory, in women who are experiencing executive functioning difficulties after having undergone a risk-reducing bilateral salpingo-oophorectomy (RRSO). This study involves magnetic resonance imaging (MRI) to see how LDX affects brain chemistry while undergoing two 6-week trials of the study drug and placebo capsules.

Individuals wishing to participate in this study are medically healthy women between the ages of 35-58 years old who have undergone a risk-reducing bilateral salpingo-oophorectomy (RRSO) within the previous 15 years. Participants must have been premenopausal before undergoing RRSO (meaning they were having regular periods). They also must not have undergone radiation or chemotherapy in the past year.

Furthermore, participants must not suffer from a mental illness, including Attention Deficit Hyperactivity Disorder (ADHD), and must not have a recent history of drug abuse. Additionally, participants must not suffer from a fear of small, enclosed spaces (claustrophobia), and not have any implanted medical devices such as a pacemaker, orthodontic braces, or shrapnel. They must not have a history of seizures, uncontrolled hypertension or known renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Age 35-58;
* Have undergone risk-reducing bilateral salpingo-oophorectomy (RRSO) within the previous 15 years AND were premenopausal at the time of RRSO;
* Score of ≥ 20 on the Brown Attention Deficit Disorder Scale (BADDS);
* Onset of executive function difficulties occurred post RRSO;
* Clean urine drug screen (nicotine and marijuana are permissible);
* Are fluent in written and spoken English;
* Are able to give written informed consent (obtained at screening visit);
* Have a high school diploma or equivalent degree (i.e., GED), as per subject report;
* If using aromatase inhibitors or tamoxifen: Must have been on a stable dose for at least 6 months;
* If completing visits remotely: Must have access to a telecommunications application (i.e., Skype), email, scanner/fax machine, and a private area that enables the protection of participant confidentiality.

Exclusion criteria:

* Current, untreated psychiatric disorder;
* Substance use disorder within the previous 3 years;
* Lifetime history of ADHD or psychotic disorder including bipolar disorder, schizoaffective disorder, and schizophrenia;
* Lifetime history of stimulant abuse or dependence;
* Regular use of psychotropic medications except selective serotonin reuptake inhibitors (SSRI), serotonin noradrenergic reuptake inhibitors (SNRI), bupropion, zolpidem, gabapentin, or buspirone;
* Chemotherapy within the past year;
* Previous history of sensitivity or adverse reaction to lisdexamfetamine (LDX);
* History of seizures or unstable medical condition;
* Known heart disease or clinically significant abnormal electrocardiogram during screening as determined by the study MD;
* Uncontrolled hypertension;
* Presence of a metallic implant contraindicative to scanning at the 7T level;
* Claustrophobia.
* Consistent systolic blood pressure of >145mm Hg or diastolic blood pressure >90 mm Hg after three readings at time of screening;
* Known renal impairment and End Stage Renal Disease (ESRD).

Ages: 35 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Neill Epperson, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- 3535 Market Street, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shanmugan S, Loughead J, Nanga RP, Elliott M, Hariharan H, Appleby D, Kim D, Ruparel K, Reddy R, Brown TE, Epperson CN. Lisdexamfetamine Effects on Executive Activation and Neurochemistry in Menopausal Women with Executive Function Difficulties. Neuropsychopharmacology. 2017 Jan;42(2):437-445. doi: 10.1038/npp.2016.162. Epub 2016 Aug 23. PMID 27550732
- [Background] Epperson CN, Shanmugan S, Kim DR, Mathews S, Czarkowski KA, Bradley J, Appleby DH, Iannelli C, Sammel MD, Brown TE. New onset executive function difficulties at menopause: a possible role for lisdexamfetamine. Psychopharmacology (Berl). 2015 Aug;232(16):3091-100. doi: 10.1007/s00213-015-3953-7. Epub 2015 Jun 11. PMID 26063677
- [Result] Brown, T. E. 1996. Brown attention deficit disorder scales for adolescents and adults, San Antonio, TX: The Psychological Corporation.
- See also: Research at the Penn Center for Women's Behavioral Wellness — http://www.med.upenn.edu/womenswellness/studies.html

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (6 Weeks)
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo, Then Lisdexamfetamine
Started | 36 | 33
Completed | 33 | 30
Not Completed | 3 | 3
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (2 Weeks)
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo, Then Lisdexamfetamine
Started | 33 | 30
Completed | 29 | 29
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 2 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo, Then Lisdexamfetamine
Started | 29 | 29
Completed | 28 | 29
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo, Then Lisdexamfetamine | Total
Number analyzed (Participants) | 36 | 33 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (5.4) | 47.3 (5.8) | 47.0 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 32 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Brown Attention Deficit Disorder Scale (BADDS) Change Score (End of Trial Minus Baseline).
Description: The Brown Attention Deficit Disorder Scale (BADDS) (Brown, 1996) is a 40-item questionnaire that assesses five subscales of executive functioning. For each item in the questionnaire, participants reported the extent to which it had been a problem over the last six months (0 = never, 1 = once a week or less, 2 = twice a week, or 3 = almost daily). Total BADDS scores can range from 0-120, with higher scores indicating more self-reported difficulties with executive functioning. Outcome measures are reported as change scores for end of trial (6 weeks) minus baseline.
Time Frame: Outcome measure change score represents end of trial (6 weeks) minus baseline.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Lisdexamfetamine (Per Intervention): Participants who received Lisdexamfetamine (20-60mg/d) in the first 6 weeks or last 6 weeks of the study.
- Placebo (Per Intervention): Participants who received placebo (1 sugar pill and will increase up to 3 pills after 4 weeks) in either the first 6 weeks or last six weeks of the study.
Arm/Group | Lisdexamfetamine (Per Intervention) | Placebo (Per Intervention)
Number analyzed (Participants) | 57 | 57
score on a scale | -19.68 [-23.17 to -16.18] | -4.31 [-7.84 to -0.78]

2. Secondary Outcome: Brain Activation (Glutamate Contrast)
Description: To measure the effects of Lisdexamfetamine on objective report of executive function difficulties proton magnetic resonance spectroscopy (1H-MRS) was utilized to assess the relative importance of dorsolateral prefrontal cortex (DLPFC) glutamate (Glut) contrast levels during working memory task performance. Measurement of glutamate contrast range from 0 to 15% with higher levels associated with optimal performance. Glutamate contrast is calculated by: GluCEST contrast (%) = [(Msat(-3ppm) - Msat(+3ppm))/Msat(-3ppm)]*100.
Time Frame: 6 weeks
Population: In response to the COVID -19 pandemic baseline neuroimaging data was only collected and analyzed on a subset of study participant (n=14).
Measure: Mean (Standard Deviation); unit: percentage of Glutmate Contrast
Groups:
- Lisdexamfetamine (Per Intervention): Participants who received Lisdexamfetamine (20-60mg/d) in the first six weeks or last six weeks of the study.
- Placebo (Per Intervention): Participants who received placebo (1 sugar pill and will increase up to 3 pills after 4 weeks) in either the first six weeks or last six weeks of the study.
Arm/Group | Lisdexamfetamine (Per Intervention) | Placebo (Per Intervention)
Number analyzed (Participants) | 14 | 14
percentage of Glutmate Contrast | 8.4 (1.03) | 8.91 (.86)

3. Secondary Outcome: Brain Activation (BOLD Percent Signal Change)
Description: To measure the effects of Lisdexamfetamine on objective report of executive function difficulties functional magnetic resonance imaging (fMRI) were utilized to assess the relative importance of dorsolateral prefrontal cortex (DLPFC) blood oxygen dependent (BOLD) signals during working memory task performance and the effect of LDX on the executive system activation. Measurement of BOLD perecent signal change range is 0 to 2%. Percent signal change is the difference in fMRI signal between the baseline condition (B) and the task condition (T) and calculated here as: percent signal change = (T-B)/B×100%. Higher percent signal change in the DLPFC is generally associated with better executive function.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Lisdexamfetamine (Per Intervention) | Placebo (Per Intervention)
Number analyzed (Participants) | 14 | 14
percentage of signal change | .42 (.229) | .21 (.223)

ADVERSE EVENTS:
Time Frame: 6 months
Description: We collected and reported all untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Lisdexamfetamine, 20 mg: Reporting AEs experienced for all participants who were exposed to Lisdexamfetamine at 20 mg. In total, 64 participants were exposed to 20mg of the drug (all participants who were exposed to LDX are included in this grouping). All AEs reported while on the 20mg dose are listed below.
  During active study participation, Participants had a 50% chance of receiving the active study medication during trial A. They began at 20 mg/d and increased up to 40 mg after 1 week and then up to 60 mg/d after 4 weeks, if well tolerated. Total time on the study drug is up to 6 weeks.
  Lisdexamfetamine: Stimulant medications are used to reduce interruptive behavior, fidgeting, and other hyperactive symptoms, as well as help a person finish tasks and improve his or her relationships for adults who have ADHD. Please note that the FDA has not approved the use of Vyvanse® for the treatment of memory and concentration difficulties related to medically induced menopause.
- Lisdexamfetamine, 40 mg: Reporting AEs experienced for all participants who were exposed to Lisdexamfetamine at 40 mg. In total, 59 participants were exposed to 40mg of the drug (5 people remained on 20mg for the duration of their trial and are not included in the 40mg or 60mg groupings). All AEs reported while on the 40mg dose are listed below.
  During active study participation, Participants had a 50% chance of receiving the active study medication during trial A. They began at 20 mg/d and increased up to 40 mg after 1 week and then up to 60 mg/d after 4 weeks, if well tolerated. Total time on the study drug is up to 6 weeks.
  Lisdexamfetamine: Stimulant medications are used to reduce interruptive behavior, fidgeting, and other hyperactive symptoms, as well as help a person finish tasks and improve his or her relationships for adults who have ADHD. Please note that the FDA has not approved the use of Vyvanse® for the treatment of memory and concentration difficulties related to medically induced menopause.
- Lisdexamfetamine, 60 mg: Reporting AEs experienced for all participants who were exposed to Lisdexamfetamine at 60 mg. In total, 43 participants were exposed to 60mg of the drug (16 people remained at 40mg, but did not increase to 60mg and therefore are not included in this 60mg grouping). All AEs reported while on the 60mg dose are listed below.
  During active study participation, Participants had a 50% chance of receiving the active study medication during trial A. They began at 20 mg/d and increased up to 40 mg after 1 week and then up to 60 mg/d after 4 weeks, if well tolerated. Total time on the study drug is up to 6 weeks.
  Lisdexamfetamine: Stimulant medications are used to reduce interruptive behavior, fidgeting, and other hyperactive symptoms, as well as help a person finish tasks and improve his or her relationships for adults who have ADHD. Please note that the FDA has not approved the use of Vyvanse® for the treatment of memory and concentration difficulties related to medically induced menopause.
- Placebo: Reporting AEs experienced for all participants who were exposed to placebo capsules. In total, 58 participants were exposed to the placebo. All AEs reported while on placebo are listed below.
  Participants will have a 50% chance of receiving the placebo for this study. They will begin with 1 sugar pill and will increase up to 3 pills after 4 weeks. Maximum time for taking the placebo is 6 weeks.
  Placebo oral capsule: The placebo capsule will be filled with microcellulose.
Arm/Group | Lisdexamfetamine, 20 mg | Lisdexamfetamine, 40 mg | Lisdexamfetamine, 60 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/59 | 0/43 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/59 | 0/43 | 0/58
Other Adverse Events (participants affected / at risk) | 2/64 | 3/59 | 12/43 | 4/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine, 20 mg (N=64) | Lisdexamfetamine, 40 mg (N=59) | Lisdexamfetamine, 60 mg (N=43) | Placebo (N=58)
Change in Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 9 (9) | 1 (1)
Difficulty falling or staying asleep (General disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Dizziness/Disorientation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 2 (2) | 9 (9) | 0 (0)
mild to moderate headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) — mild to moderate headache
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Increased blood pressure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Blood pressure increased above normal reading
Drowsiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea/Gas (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Jitters (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Soreness/Tingling Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 3 (4) | 2 (2)
Increased Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03187353/Prot_SAP_000.pdf